CLINICAL TRIAL: NCT01952288
Title: Simvastatin: Proof-of-Concept for Prevention of Neurodegeneration in Mild TBI
Brief Title: Simvastatin for mTBI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: B1195-I
Record Dates: First submitted 2013-09-24; First posted 2013-09-27 (Estimated); Results first posted 2021-12-15 (Actual); Last update posted 2021-12-15 (Actual); Status verified 2021-11

CONDITIONS: TBI-Traumatic Brain Injury
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Simvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- simvastatin (Experimental): simvastatin 40 mg/day
  Interventions: Drug: simvastatin
- placebo (Placebo Comparator): placebo
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: simvastatin — simvastatin 40 mg/day for 12 months
  Other Names: Zocor
  Arms: simvastatin
Drug: Placebo Oral Tablet — placebo comparator
  Arms: placebo

SUMMARY:
Study of simvastatin in Iraq/Afghanistan Veterans with multiple blast exposure and mTBI. The study will measure substances in cerebrospinal fluid (CSF) that are related to dementing disorders.

DETAILED DESCRIPTION:
Many Iraq and Afghanistan Veterans have experienced repetitive blast exposure mild traumatic brain injury (mTBI) with persistent cognitive, emotional, and neurological postconcussive symptoms. There is an urgent need to develop effective treatments to reduce both the intensity of these Veterans' current symptoms as well as their potential long-term risks for developing neurodegenerative dementing disorders related to repetitive mTBI: chronic traumatic encephalopathy (CTE) and Alzheimer's disease (AD). Converging evidence suggests that statins may possess neuroprotective effects against pathologic processes related to tau protein metabolism that appear to be a common feature of CTE, AD, and other neurodegenerative sequelae of repetitive mTBI.

The investigators propose a 12-month, double-blind, randomized, active-drug-controlled trial to establish proof-of-concept for use of simvastatin (40 mg/d) for decreasing CSF biomarkers of neurodegeneration and increasing CSF neurotrophins in 120 Iraq and Afghanistan Veterans with repetitive blast trauma mTBI.

ELIGIBILITY:
Inclusion Criteria:

* Males and females ages 21-50 years.
* Documented hazardous duty in Iraq and or Afghanistan with the U.S. Armed Forces.
* Exposure to one or more blast trauma events resulting in mTBI according to American Congress of Rehabilitation Medicine (ACRM) criteria.
* More than 6 months since last blast trauma exposure
* Ability to complete psychometric and other clinical assessments in English (i.e., adequate English language skills, vision and hearing).
* elevated cholesterol levels, i.e. total cholesterol >200 and/or LDL >130. This would generally prompt the initiation of a lipid-lowering agent as standard care in the general medical community.
* No use of statins during the previous year and no recent (past 4 weeks) use of other lipid-lowering drugs (e.g., fibrates, niacin > 500mg/d, or high dose omega-3 fatty acids) preceding randomization.
* No clinically significant laboratory abnormalities (electrolytes, glucose, carbon dioxide, blood urea nitrogen (BUN), creatinine, vitamin B12, folate, albumin, thyroid stimulating hormone).
* Platelet count > 100,000/mm2.
* Body Mass Index (BMI) between 18 and 36 inclusive

Exclusion Criteria:

* History of head trauma with loss of consciousness (LOC)>30 minutes, or with a penetrating head wound, or with moderate to severe memory or other cognitive impairment.
* Neurological disorders: multiple sclerosis, epilepsy, stroke, Parkinson's disease (PD), other degenerative Central Nervous System (CNS) disorders, or neuropathy with radicular involvement.
* Acute or chronic major psychiatric disorders: schizophrenia, bipolar disorder or severe major depressive disorder, or severe anxiety disorder except PTSD and panic disorder (PTSD and depressive symptoms are common co-morbid conditions for combat mTBI and a subset of these patients have symptoms consistent with panic disorder as well).
* Use of illegal drugs; alcohol abuse within the past 6 months.
* Poorly controlled hypertension, heart failure, coronary heart disease, peripheral artery disease, carotid artery disease, diabetes mellitus, pulmonary disease with hypoxia or hypercapnia, significant hepatic disease or hepatitis C seropositivity, renal failure, treatment for cancer, HIV positive, active infectious disease or presence of abdominal aortic aneurysm.
* Contraindications to lumbar puncture (LP) (e.g., spinal cord injury; deformity, severe disease or infection in the region of the lumbosacral spine; bleeding tendency, use of anticoagulant medications, or platelet count <100,000/mm2).
* Receiving medication in an investigational drug study.
* Exclusionary medications (used in the 4 weeks prior to screening):
* Fibrates and niacin due to increased risk for myopathy in combination with statins;
* Potential drug-drug interactions with statins via effects on CYP3A4: itraconazole, ketoconazole, erythromycin, clarithromycin, HIV protease inhibitors, nefazodone, amiodarone, cyclosporine, isoniazid, quinidine, or large quantities of grapefruit juice (>1 quart daily);
* Selected CNS-acting medications: antipsychotics, anti-Parkinson's disease medications and CNS stimulants
* Other medications affecting coagulation and/or inflammation: coumadin, potent anti-inflammatory medications (hydrocortisone, methotrexate or other potent immune-modulating medications), and anti-HIV medications.
* All female subjects of childbearing potential will undergo a urine pregnancy test at every subject visit; subjects with positive pregnancy test results will be excluded. In addition, all female subjects of childbearing potential will be required to use a reliable method of contraception throughout the duration of the study.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2013-09-16 (Actual); Primary Completion 2017-06-20 (Actual); Study Completion 2017-06-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elaine R Peskind, MD, Principal Investigator — VA Puget Sound Health Care System Seattle Division, Seattle, WA
Locations (1):
- VA Puget Sound Health Care System Seattle Division, Seattle, WA, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Riekse RG, Li G, Petrie EC, Leverenz JB, Vavrek D, Vuletic S, Albers JJ, Montine TJ, Lee VM, Lee M, Seubert P, Galasko D, Schellenberg GD, Hazzard WR, Peskind ER. Effect of statins on Alzheimer's disease biomarkers in cerebrospinal fluid. J Alzheimers Dis. 2006 Dec;10(4):399-406. doi: 10.3233/jad-2006-10408. PMID 17183151
- [Background] Li G, Mayer CL, Morelli D, Millard SP, Raskind WH, Petrie EC, Cherrier M, Fagan AM, Raskind MA, Peskind ER. Effect of simvastatin on CSF Alzheimer disease biomarkers in cognitively normal adults. Neurology. 2017 Sep 19;89(12):1251-1255. doi: 10.1212/WNL.0000000000004392. Epub 2017 Aug 18. PMID 28821686

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Simvastatin | Placebo
Started | 3 | 2
Completed | 3 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Simvastatin | Placebo | Total
Number analyzed (Participants) | 3 | 2 | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 2 | 5
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 3 | 2 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 2 | 5
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 2 | 1 | 3
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Cerebrospinal Fluid (CSF) T-tau Concentration
Description: Change in CSF total tau concentration from baseline to 12 months of study drug treatment
Time Frame: baseline, 12 months
Measure: Mean (Standard Error); unit: pg/ml
Arm/Group | Simvastatin | Placebo
Number analyzed (Participants) | 3 | 2
pg/ml | 24 (20) | 33.5 (17)

2. Primary Outcome: Cerebrospinal Fluid (CSF) P-tau 181 Concentration
Description: Change in CSF p-tau 181 concentration from baseline to 12 months of study drug treatment
Time Frame: baseline, 12 months
Measure: Mean (Standard Error); unit: pg/ml
Arm/Group | Simvastatin | Placebo
Number analyzed (Participants) | 3 | 2
pg/ml | 3.1 (2) | 1.6 (1.4)

3. Secondary Outcome: CSF Abeta 1-40 Concentration
Description: change in CSF abeta 1-40 concentration from baseline to 12 months of study drug treatment
Time Frame: baseline, 12 months
Measure: Mean (Standard Error); unit: pg/ml
Arm/Group | Simvastatin | Placebo
Number analyzed (Participants) | 3 | 2
pg/ml | 753 (363) | 953 (710)

4. Secondary Outcome: CSF Abeta 1-42 Concentration
Description: change in CSF abeta 1-42 concentration from baseline to 12 months of study drug treatment
Time Frame: baseline, 12 months
Measure: Mean (Standard Error); unit: pg/ml
Arm/Group | Simvastatin | Placebo
Number analyzed (Participants) | 3 | 2
pg/ml | 43 (24.5) | 82.5 (58.5)

ADVERSE EVENTS:
Time Frame: baseline through 12 months study participation
Arm/Group | Simvastatin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/2
Other Adverse Events (participants affected / at risk) | 3/3 | 2/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Simvastatin (N=3) | Placebo (N=2)
Upper Respiratory Infection (Infections and infestations) | 2 (2) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 1 (2)
Increased Confusion (Nervous system disorders) | 1 (1) | 0 (0)
nasal congestion (General disorders) | 1 (1) | 0 (0)
Tonsillitis (Infections and infestations) | 1 (1) | 0 (0)
Sciatica (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
night sweats (General disorders) | 0 (0) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Shoulder pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Recruitment difficulties (persons with normal cholesterol levels were not interested in taking statins) led to not enrolling sufficient numbers of participants to achieve target power.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-11-16): https://cdn.clinicaltrials.gov/large-docs/88/NCT01952288/Prot_SAP_000.pdf